CLINICAL TRIAL: NCT05745324
Title: The Effect of Scaling and Root Planing on Gingival Crevicular Fluid and Salivary Levels of Inflammatory Biomarkers Among Electronic Nicotine Delivery Systems User, Smokers and Non-Smokers
Brief Title: The Effect of Scaling and Root Planing on Oral Inflammatory Biomarkers Among E-cig Users and Non-smokers
Acronym: ENDS-SRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr Jagan K Baskaradoss, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VDR/ED/14
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Diseases; Smoking
Keywords: electronic cigarettes
MeSH Terms: conditions — Periodontal Diseases; Smoking; Vaping | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators, care providers and outcome assessors would be blinded to the smoking status of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smoker vs Nonsmokers (Experimental): SRP would be performed for Smokers (ENDS and conventional cigarette) and Nonsmokers and their inflammatory biomarkers would be assessed.
  Interventions: Procedure: Scaling and root planing
- ENDS users and Nonsmokers (Experimental): SRP would be performed for ENDS users and Nonsmokers and their inflammatory biomarkers would be assessed.
  Interventions: Procedure: Scaling and root planing
- Smokers with periodontitis and Nonsmokers (Experimental): SRP would be performed for Smokers with periodontitis and health nonsmokers and their inflammatory biomarkers would be assessed.
  Interventions: Procedure: Scaling and root planing
- Smokers with periodontitis and Nonsmokers with periodontitis (Experimental): SRP would be performed for Smokers and Nonsmokers with periodontitis and their inflammatory biomarkers would be assessed.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — SRP is cleaning the sub gingival and supra gingival plaque and calculus from the teeth

SUMMARY:
Background/Aim: There are no studies that have compared the gingival crevicular fluid (GCF) levels of IL-1β in non-smokers (NS) and electronic nicotine delivery system (ENDS)-users before and after scaling and root planing (SRP) in patients with gingivitis. The aim of the present study is to compare the effect of scaling and root planing on the expression of IL-1β in the GCF among ENDS-users and NS clinically.

Methods: Self-reported current ENDS users and NS would be included. A questionnaire would be used to collect demographic data. All patients would undergo SRP. Clinical measures, periodontal parameters [probing depth (PD), plaque index (PI), and bleeding on probing (BOP)], and GCF IL-1β would be measured at baseline. At 1-week (T1) and 3 weeks (T2) of follow-up, periodontal parameters and GCF IL-1β levels would be re-assessed.

DETAILED DESCRIPTION:
2.1. Ethical approval Ethical approval was obtained from the Ethics Committee of Health Sciences Center at Kuwait University. All volunteering individuals were requested to read and sign a consent form written in simple English and Arabic.

2.2. Study Area/Setting The present longitudinal study was conducted between November 2021 and September 2022 at the Kuwait University Dental Center (KUDC). The study participants were regular patients attending the KUDC and the sampling design was convenience sampling.

2.3. Selection Criteria The inclusion criteria: ENDS-users, non-smokers, age (18-25), gender (men), periodontal health status (gingivitis), having minimum number of 20 teeth, and medically healthy. The exclusion criteria: Patients who did scaling and root planing in the past 3 months, T-cigs smokers, and dual smokers.

2.4. Data Collection Methods, Instrument Used, Measurements A standardized questionnaire including a consent form was used to gather information regarding gender, age (in years), nationality, marital status, highest level of education, oral hygiene status, last dental visit, last time that scaling and root planing was done, smoking status, type of smoked product, duration of ENDS usage (in years), frequency of ENDS usage per day, number of ENDS puffs taken per session, family smoking history, exposure to secondhand smoke, general health status, and attitude towards smoking.

2.5. Blinding

2.6. Study Participants Twenty current ENDS-users and eighteen NS were recruited to participate in this study. All participants were requested to refrain from eating and using any oral hygiene method for at least 3 hours prior to their visit.

2.7. Sample Collection For screening of subjects for their use of tobacco products, saliva was collected and tested for the content of nicotine using chairside test kits (NicAlert, Confirm Bioscience, CA, USA). Unstimulated saliva (UWS) was collected before clinical assessment using non-invasive techniques. Prior to salivary and GCF samples collection, each participant's vital signs were measured and recorded. The participants were asked to rinse their mouth with water before a baseline salivary sample is collected to measure cotinine levels. Each participant was asked to collect saliva passively in their mouth and expectorate in a tube every one minute until three millimeters of saliva is collected. The tubes were then stored at -80°C. After that, GCF samples were collected using filter paper strips. GCF will be sampled from four sites at fully erupted, caries-free permanent molars (mesiobuccal and distobuccal of each molar) with gingival index (GI) score of 2 or 3 for gingivitis group. Scaling and root planing was provided for each participant and saliva and GCF samples were obtained in the same manner explained previously after one week and three weeks.

2.8. Power Analysis Power analysis was determined using a computer software (nQuery Advisor 6.0, Statistical Solutions, Saugas, MA., USA) with an alpha and effect size of 0.05 and 0.3, respectively. Sample size estimation was based on the presumption that a mean difference of 1 mm in clinical AL and PD should be detected at a significance-level of 0.05 and a desired study power of at least 80%. It was estimated that a sample size of at least 20 patients/group would achieve 95% study power with a 0.05 two-sided significance-level.

2.9. Analysis of Cotinine and IL-1β in GCF Saliva levels of cotinine was measured to determine the electronic cigarettes status using a high sensitivity, quantitative enzyme immunoassay (ELISA) kit. Then, IL-1β GCF levels was analyzed using commercially available ELISA kit. The difference in the levels of the biomarker before and after the intervention will provide an insight of the soft tissue response to the treatment. This will show the deleterious effect of electronic nicotine delivery systems on the soft tissue response to therapy.

2.10. Clinical Examination In all patients, Löe & Silness gingival index (GI)(Löe and Silness 1963) and Silness & Löe plaque index (PI)(Silness and Löe 1964) were recorded.

2.11. Statistical Analysis Statistical analyses was done using SPSS software (SPSS Version 26, Chicago, IL., USA).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria: ENDS-users, cigarette smokers, non-smokers, age (18-60), gender (men), periodontal health status (gingivitis/periodontitis), having minimum number of 20 teeth, and medically healthy.

Exclusion Criteria:

* The exclusion criteria: Patients who did scaling and root planing in the past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 3 months
  Level of gingival attachment would be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Kuwait City, Kuwait

REFERENCES:
- [Derived] Alkhalifah AB, Alfuraih NT, Joseph B, Baskaradoss JK. Effect of scaling on levels of interleukin 1-beta and clinical periodontal parameters among e-cigarette users and non-smokers: A prospective study. Tob Induc Dis. 2024 Jul 10;22:10.18332/tid/189552. doi: 10.18332/tid/189552. eCollection 2024. PMID 38988743